CLINICAL TRIAL: NCT05099302
Title: The Effect of Cartoons Watched Before Surgery on Children's Fear Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Sonay Turkmen, Prof.Dr (Other)
Responsible Party: Sponsor-Investigator, Ayse Sonay Turkmen, Prof.Dr, Assoc.Prof., Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: CARTOONS1
Record Dates: First submitted 2021-09-28; First posted 2021-10-29 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2021-10

CONDITIONS: Preoperative; Cartoon; Fear; Appendectomy; Tonsillectomy
Keywords: preoperative period; watching cartoons; fear in children

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cartoon group (Experimental): In the research, the group whose fear was tried to be reduced by watching cartoons
  Interventions: Other: divert attention
- control group (No Intervention): The group whose change in the process was monitored without any intervention in the research

INTERVENTIONS:
Other: divert attention — In order to reduce the fears of the children who came to the waiting room before the operation, they watched cartoons and their attention was diverted to another point.
  Arms: cartoon group

SUMMARY:
This study was conducted as a randomized controlled experimental study to determine the effect of cartoon in reducing pre-operative fear in children aged 4-10 years who came to the operating room. The data of the study were obtained from children between 4-10 years old who came to Mersin University Hospital Operating Room Unit between 1 July and 30 August 2020. The sample size was determined as a total of 116 children, including 58 children for each group. "Observation Form, Children's Fear Scale (CFS), Tablet Computer, Stopwatch" was used for data collection. The data were evaluated using percentage, mean, standard deviation, chi-square, t test, Anova and Tukey advanced analysis test.

Cartoons group; When the children came to the operating room waiting room, the first stopwatch was started as soon as they entered the room to determine the length of stay in the waiting room, and it was turned off while they were entering the operating room with the anesthesiologist. Thus, the total length of stay in the room was determined and recorded. The second stopwatch was started as soon as the child began to cry, and was turned off when the crying stopped. Thus, the crying time of each child was also evaluated. After each parent signed the Informed Consent Form, the Interview and Observation Form was filled. Then the child's heart rate was measured and recorded. The child's fear level was evaluated separately by the child, parent and observer via CFS and recorded in the data collection form. After the initial assessment was completed, the child was asked if he wanted to watch cartoons. "Snow Queen" for girls who want to watch cartoons and "Spider-Man" cartoons for boys started to be watched by tablet. The period of watching cartoons lasted until the child left the waiting room. The heart rate was measured just before the child left the waiting room at the time of surgery. The level of fear was evaluated separately by the child, parent and observer via CFS and recorded in the form. Then, the child was taken to the operating room with the anesthesiologist and observer. Parents are separated from their children in the waiting room. After the child who came to the operating room was taken to the operating table, the pulse rate and the level of fear were evaluated and recorded by the observer via CFS.

Control group: All processing steps were carried out similarly to the cartoon group. In this group, the option of playing toys was offered instead of cartoons.

DETAILED DESCRIPTION:
The research will be carried out in the Operating Room Unit of X University Hospital. There are 20 surgical specialists, eight anesthesiologists, 35 nurses, 25 anesthesia technicians, 30 support personnel, and personnel working in 13 different areas (such as secretary, consumables warehouse manager) in the operating room unit. The personnel working in the unit working in shifts work in shifts between 08.00-16.00, 16.00-08.00 and 16.00-24.00. There are 16 operating rooms in total in the operating room unit. Apart from these rooms, there are pre-operative patient waiting room, pre-operative pediatric waiting room and postoperative patient/children's rooms. There are also rest rooms for the personnel working in the operating room and a 10-bed reanimation unit. The pre-operative pediatric waiting room is located at the patient admission entrance of the operating room and is not a sterile area. It has an average size of 40 m2 and includes a television, two beds, two armchairs and toys. There are cartoon characters and pictures on the walls of the waiting room. Before the operation, children spend an average of 5-20 minutes in the children's waiting room after the operation. is brought first. After the necessary procedures are performed by the preop nurse, the child is taken to the operating room in the presence of an anesthesiologist and anesthesiologist.

The sample size was calculated with 95% power, with 10% difference at 0.05 significance level, taking into account the known score (4.53 ± 3.23) with the G*Power 3.1.5 program. The sample size was determined as 58 children for each group. A total of 116 children were not reached. At the end of the study, Post Hoc power analysis will also be carried out in order to determine the adequacy of the number of children included in the study, and if 95% power is reached, the data collection process will be terminated.

Randomization of control and study groups; The status of the children to be included in the study in the control or study group will be determined by using "stratification and randomization methods with blocks". In the literature, it has been reported that among the factors affecting the fear and anxiety experienced by children in interventional procedures, variables such as age, gender and fear of interventional procedure are included. Accordingly, block randomization will be applied by stratifying the children as "girl and boy" for the gender variable and "4 years, 5 years and 6 years and over" for the age variable. 58 children will be included in each of the research groups. During the data collection process, each child and his/her family will be taken to the operating room waiting room one by one. This will prevent children from meeting each other.

ELIGIBILITY:
Inclusion Criteria:

the child;

* Age between 4-10 years
* Children's perception level to evaluate the scale of fear
* The child does not have any physical or mental illness
* The child's ability to communicate and be open to communication
* The child does not have a hearing, speech or vision problem
* The child does not have a long-term illness
* The child and his parents agree to participate in the study.

Exclusion Criteria:

* The child is less than 4 years old or over 10 years old,
* The presence of any chronic disease, physical or mental illness that may affect the child's fear state
* Child or family refusal to participate in the study

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Fear Scores | 15 minutes
  Changes from Baseline in Visual Analogue Scale Fear Scores in Children with Operation-Related Fear Evaluated by CFS at Entrance to the Operating Room, Leaving the Waiting Room, and at the Operating Table.
Heart Rate | 15 minutes
  Changes from Baseline in heart rate in Children with Operation-Related at Entrance to the Operating Room, Leaving the Waiting Room, and at the Operating Table.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KaramanogluMehmetbeyU, Karaman, Turkey
  - Karamanoglu Mehmetbey University, Karaman

IPD SHARING:
Plan to Share IPD: No